CLINICAL TRIAL: NCT06315712
Title: Effects of Adding Inspiratory Muscle Training to Pulmonary Rehabilitation Program in Adults With Burn Injuries: A Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training in Burned Adults
Acronym: Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Applied Medical Sciences, Qassim University, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 004201
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Burn Injuries
MeSH Terms: conditions — Burns | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle training group (Experimental): Received inspiratory muscle training plus pulmonary rehabilitation program. Powerbreathe device was used for the exercise of the inspiratory muscle strength. Strengthening the inspiratory muscles with the Powerbreathe is similar to weightlifting to strengthen other muscles in the body.
  Interventions: Other: inspiratory exercise; Other: Pulmonary rehabilitation
- Pulmonary rehabilitation group (Experimental): Received pulmonary rehabilitation program for five sessions per week for 8 weeks. Four resistive exercises, aerobic exercise, and deep breathing exercises, aerobic conditioning exercises on the treadmill. All exercises were performed using variable resistance machines.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: inspiratory exercise — The training consisted of 6 sets of 30 breaths per day, divided into 2 sessions per day. A one-minute rest interval between each set. Training was prescribed 5 days a week for 8 weeks
  Other Names: inspiratory muscle training
  Arms: Respiratory muscle training group
Other: Pulmonary rehabilitation — Four resistive exercises, aerobic exercise, and deep breathing exercises, five sessions per week for 8 weeks
  Other Names: Resistance exercise

SUMMARY:
The study outlines burn injury impact, emphasizes need for long-term rehabilitation. Study assesses inspiratory muscle training efficacy in improving respiratory strength, lung function, and exercise capacity in adult burn patients.

DETAILED DESCRIPTION:
The study aimed to evaluate the effectiveness of adding inspiratory muscle training to pulmonary rehabilitation in adult burn patients. Fifty-two participants were randomly assigned to either inspiratory muscle training plus pulmonary rehabilitation or pulmonary rehabilitation alone for 8 weeks. Inspiratory muscle training consisted of using a Powerbreathe device for inspiratory muscle strengthening.

ELIGIBILITY:
Inclusion Criteria:

* Burn-injured adults aged 20-49.
* Admitted to the clinic after acute treatment.
* Recovering from burns affecting at least 20% total body surface area.
* Partial or full-thickness burns.

Exclusion Criteria:

* Smokers.
* had open or unhealed wounds.
* had any known neurological deficit.
* neuromuscular diseases.
* musculoskeletal deformities.
* pulmonary diseases.
* severe cardiac problems.
* inability to participate in regular exercise.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
maximal inspiratory pressure | At the beginning of intervention
  performed using an electronic respiratory pressure meter, measures inspiratory muscle strength
maximal inspiratory pressure | After 8 weeks of intervention
  performed using an electronic respiratory pressure meter, measures inspiratory muscle strength
maximal expiratory pressure | At the beginning of intervention
  performed using an electronic respiratory pressure meter, assesses expiratory muscle strength.
maximal expiratory pressure | After 8 weeks of intervention
  performed using an electronic respiratory pressure meter, assesses expiratory muscle strength.
Forced expiratory volume in 1 second | At the beginning of intervention
  performed using a spirometer
Forced expiratory volume in 1 second | After 8 weeks of intervention
  performed using a spirometer
forced vital capacity | At the beginning of intervention
  performed using a spirometer
forced vital capacity | After 8 weeks of intervention
  performed using a spirometer
Forced expiratory volume in 1 second/ forced vital capacity ratio | At the beginning of intervention
  performed using a spirometer
Forced expiratory volume in 1 second/ forced vital capacity ratio | After 8 weeks of intervention
  performed using a spirometer

SECONDARY OUTCOMES:
Functional exercise capacity | At the beginning of intervention
  assessed using the six-minute walk test
Functional exercise capacity | After 8 weeks of intervention
  assessed using the six-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: FatmaAlzahraa Kamel, PhD, Principal Investigator — Cairo University; Maged Basha, PhD, Study Chair — Qassim University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Willis CE, Grisbrook TL, Elliott CM, Wood FM, Wallman KE, Reid SL. Pulmonary function, exercise capacity and physical activity participation in adults following burn. Burns. 2011 Dec;37(8):1326-33. doi: 10.1016/j.burns.2011.03.016. Epub 2011 May 6. PMID 21530086
- [Background] Ozkal O, Topuz S, Karahan S, Erdem MM, Konan A, Yasti AC. Clinical predictors of pulmonary functions, respiratory/peripheral muscle strength and exercise capacity at discharge in adults with burn injury. Disabil Rehabil. 2021 Oct;43(20):2875-2881. doi: 10.1080/09638288.2020.1720320. Epub 2020 Jan 30. PMID 31999499
- [Result] Gittings PM, Grisbrook TL, Edgar DW, Wood FM, Wand BM, O'Connell NE. Resistance training for rehabilitation after burn injury: A systematic literature review & meta-analysis. Burns. 2018 Jun;44(4):731-751. doi: 10.1016/j.burns.2017.08.009. Epub 2017 Oct 7. PMID 29017743